CLINICAL TRIAL: NCT04505514
Title: Single Dose Intravenous Iron Isomaltoside in Combination With Oral Iron vs Oral Iron Monotherapy in Patients With Anemia After Postpartum Haemorrhage: A Single-blinded, Randomised Controlled Trial
Brief Title: Single Dose Intravenous Iron Isomaltoside in Combination With Oral Iron vs Oral Iron Monotherapy in Patients With Anemia After Postpartum Haemorrhage
Acronym: IVIronPPH
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Carolyn Yim Chue Wai, Consultant Anaesthesiologist, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020121-8204
Record Dates: First submitted 2020-07-23; First posted 2020-08-10 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Post Partum Hemorrhage; Anemia
MeSH Terms: conditions — Postpartum Hemorrhage; Anemia | interventions — iron isomaltoside 1000

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous Iron Group (Experimental)
  Interventions: Drug: Iron Isomaltoside 1000; Drug: Iberet-Folic-500
- Oral Iron Group (Active Comparator)
  Interventions: Drug: Placebo; Drug: Iberet-Folic-500

INTERVENTIONS:
Drug: Iron Isomaltoside 1000 — single dose of 1000 mg iron isomaltoside diluted in 100 ml of 0.9% sodium chloride, infused intravenously over ≥ 20 minutes.
  - infusion set will be covered for blinding
  Arms: Intravenous Iron Group
Drug: Placebo — 100 ml of 0.9% sodium chloride, infused intravenously over ≥ 20 minutes.
  - infusion set will be covered for blinding
  Arms: Oral Iron Group
Drug: Iberet-Folic-500 — once a day dose, to start 5 days after the intervention

SUMMARY:
The investigator's study is going to compare effectiveness of single dose intravenous iron in combination with oral iron versus oral iron monotherapy in correcting haemoglobin deficit, replenishing iron stores and improving clinical symptoms in women with post-partum anaemia after postpartum hemorrhage without increasing the rate of adverse outcomes.

ELIGIBILITY:
Inclusion Criteria:

* women who underwent spontaneous vaginal delivery with Post partum hemorrhage (PPH) ≥ 500ml OR women who underwent lower segment caesarean section with PPH ≥ 1000 ml
* post PPH haemoglobin level ≤ 10.0 g/dl measured within 48hrs after delivery and stabilisation & resuscitation.
* ≥ 18 years of age
* Proficient in Malaysian language or English language
* Willingness to consent for blood taking and attending follow-up at 2 weeks and 6 weeks

Exclusion Criteria:

* refused consent to participate in trial
* history of hemolytic anemia, Thalassemia , and sickle cell anemia
* women with signs of sepsis (clinical or laboratory evidence-intrapartum fever >38.5 degrees with abnormal vital signs, positive blood culture)
* clinical or laboratory evidence of hepatic or renal, cardiovascular and hemolytic abnormalities
* history of active severe acid peptic disorder, esophagitis or hiatus hernia and malabsorption syndrome.
* Severe symptoms of anemia including dyspnoea at rest, angina pectoris, syncope or transient ischemic attacks.
* history of severe asthma, eczema or other atopic allergy
* known allergy to iron
* patients with known immune or inflammatory conditions (e.g. systemic lupus erythematosus, rheumatoid arthritis).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin concentration (g/dL) | Six weeks after intervention
  To evaluate the increase in hemoglobin level
Serum iron concentration | Six weeks after intervention
  To evaluate the increase in serum iron concentration (µmol/L)
Serum ferritin concentration | six weeks after intervention
  serum ferritin levels (µg/L)

SECONDARY OUTCOMES:
General fatigue score | Six weeks after intervention
  Using the Multidimensional Fatigue Inventory (MFI) which will be answered by the participants, scores will be taken ranging from lowest 4, till the highest of 20. A higher score will indicate higher levels of fatigue.
Number of participants that had adverse effects to intravenous iron | Up to six weeks after intervention
  Any adverse effects experienced by the participant arising from the administration of intravenous iron isomaltoside will be documented and managed as per protocol.
Blood transfusion requirement | Up to six weeks after intervention
  Number of blood transfusions required after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- University of Malaya Medical Centre, Petaling Jaya, Kuala Lumpur, Malaysia